CLINICAL TRIAL: NCT01282047
Title: Multicenter, Open Label, Phase II Trial to Evaluate the Efficacy and Safety of Treatment With Lenalidomide in Kaposi Disease Associated With HIV Infection (ANRS 154/LENAKAP)
Brief Title: Lenalidomide in Kaposi Disease Associated With HIV Infection
Acronym: LENAKAP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-022898-33; ANRS 154 LENAKAP
Record Dates: First submitted 2011-01-21; First posted 2011-01-24 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: HIV Infection Associated Kaposi Disease
Keywords: Lenalidomide; Kaposi; HIV; efficacy; safety
MeSH Terms: interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide (Experimental)
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — oral course, 25 mg, day 1 to 21, per month, 7 days of wash-out each month. Duration according to initial response: 24 weeks and 12 weeks more if complete remission, 24 weeks more if partial remission or stable disease and stop in case of progression.

SUMMARY:
Lenakap : This multicenter, non randomized (single arm), open, phase II study aims to evaluated the efficacy of Lenalidomide in HIV-associated kaposi disease. Patients will be followed for 48 weeks. Measurement of primary endpoint will be at 24 weeks.

DETAILED DESCRIPTION:
Lenakap : This multicenter, non randomized (single arm), open, phase II study aims to evaluated the efficacy of Lenalidomide in HIV-associated kaposi disease. Patients will be followed for 48 weeks. Measurement of primary endpoint will be at 24 weeks.

The observation period is 48 weeks. The main criteria is evaluated at 24 weeks Inclusion period: 72 weeks from the setting-up meeting.Lenalidomide will be stopped in the case of progression and the patients will be considered as drop-out from the trial, but will be taken into account in the final analysis.

Two-steps procedure: 14 evaluable patients in the first step; if one response to treatment is observed, other patients are included up to 25 evaluable patients.

ELIGIBILITY:
Inclusion Criteria:

* Men or non childbearing (negative serum Human Chorionic Gonadotropin-hCG) non breastfeeding women who practice adequate birth control, maintained 4 weeks after stopping lenalidomide
* Age over 18 years and below 75 years
* Able and willing to give written informed consent
* Serologic documentation of HIV infection by approved tests, undetectable HIV viral load (below 50 copies/mL) independently of CD4 cell counts
* Biopsy proven symptomatic Kaposi sarcoma with at least 4 measurable cutaneous lesions
* Treatment by cART for at least 12 months, without wash out the last 6 months with undetectable HIV-RNA (below 50 copies/mL)
* History of treatment failure or relapse with 1 or more chemotherapy
* Progressive disease with need to new specific therapy
* Wash-out over 4 weeks if previous specific Kaposi sarcoma chemotherapy (8 weeks if Interferon -IFN therapy)
* Karnofsky performance status over 70%
* Social security (State Medical Assistance is not a social security scheme)
* Agree to abstain from donating blood
* Agree not to donate semen
* Agree not to share study drug with another person

Exclusion Criteria:

* Childbearing or breastfeeding (positive betaHCG serum)
* Kaposi sarcoma with only visceral locations
* Kaposi sarcoma with cardiac and/or bronchopulmonary localisations
* 2 viral loads over 50 copies/mL under Highly active antiretroviral therapy (HAART), during the last 6 months
* Opportunistic infections, uncontrolled infections
* Cardiac disease
* Castleman disease or lymphoma
* Other cancers or previous or current haematological malignancies
* Polyneuritis, grade over 2
* Association with neurotoxic drugs such as isoniazid, d4T
* Neutrophil polynuclear count below 1000/mm3 or platelets below 75000/mm3
* Life expectation under 2 months
* Creatinine clearance below or equal 50 mL/min (Cockcroft-Gault formula)
* Serum Glutamopyruvate Transferase (SGPT) or Serum Glutamooxaloacetate Transferase (SGOT) over or equal 3
* Concomitant treatment with antineoplastic drugs
* Known allergy or hypersensitivity to aspirin, to lenalidomide
* Contraindication to anticoagulant drugs
* Safeguard justice

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of treatment with Lenalidomide in progressive Kaposi disease in Human immunodeficiency virus (HIV)-infected patients receiving Combined Antiretroviral Therapy (cART). | Clinical benefit at week 24
  For all patients clinical tumour evaluation : complete clinical examination, tumour scoring according to the Aids Clinical Trials Group (ACTG) and The Physician's Global Assessment (PGA) and laboratory assessment.
  Any patient in documented progression during treatment will be withdrawn from the trial and declared to be in disease progression for the final evaluation but followed monthly like other participants. Such patients will be treated under the physician's responsability.

SECONDARY OUTCOMES:
To estimate the safety of lenalidomide | From Week 0 to Week 48
  All patients that have started one dose of active treatment will be included in the analysis of safety.
  Adverse event will be described precisely for each patient and for each event according to ANRS adverse events criteria. A descriptive analysis of each laboratory result and vital signs will be provided.
To estimate the time to the response and the duration of the response | From Week 0 to Week 48
To evaluate the efficacy of treatment at 48 weeks | Week 48
  The analysis of efficacy will determine the proportion of patients with objective response according to the Physical Global Assessment (PGA) score at week 24 and using ACTG criteria for Kaposi.
To evaluate the efficacy using ACTG criteria | From Week 0 to Week 48
To evaluate the survival and the survival with no progression | From Week 0 to Week 48
To describe the evolution of virologic and immunological parameters | From Week 0 to Week 48
  To describe the evolution of virologic and immunological parameters:
  CD4 and CD8 cell counts, Plasma HIV and HHV8 loads
To estimate the safety of lenalidomide | From Week 0 to Week 48
  All patients that have started one dose of active treatment will be included in the analysis of safety.
  Adverse event will be described precisely for each patient and for each event according to French AIDS Agency (ANRS) adverse events criteria. A descriptive analysis of each laboratory result and vital signs will be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Martinez, MD, PhD, Principal Investigator — APHP, Hopital Beclere, Clamart France; Dominique Costagliola, PhD, Study Director — U943 INSERM and Université Pierre et Marie Curie
Locations (1):
- Valerie Martinez, Clamart, France, France

REFERENCES:
- [Derived] Pourcher V, Desnoyer A, Assoumou L, Lebbe C, Curjol A, Marcelin AG, Cardon F, Gibowski S, Salmon D, Chennebault JM, Poizot-Martin I, Peytavin G, Boue F, Costagliola D. Phase II Trial of Lenalidomide in HIV-Infected Patients with Previously Treated Kaposi's Sarcoma: Results of the ANRS 154 Lenakap Trial. AIDS Res Hum Retroviruses. 2017 Jan;33(1):1-10. doi: 10.1089/AID.2016.0069. Epub 2016 Sep 7. PMID 27405442
- See also: Related Info — http://www.anrs.fr